CLINICAL TRIAL: NCT03830567
Title: Pharmacists Expand Access to Reproductive Healthcare: Reducing Unintended Pregnancy Through Pharmacist Prescription of Contraception
Brief Title: Pharmacists Expand Access to Reproductive heaLthcare
Acronym: PEARL
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Laura and John Arnold Foundation (Other)
Responsible Party: Principal Investigator, Maria Rodriguez, MD, MPH, Associate Professor, Oregon Health and Science University
Other Study IDs: OHSU IRB 16158
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Contraception
Keywords: Hormonal Contraception; Birth Control; Pharmacists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pharmacist prescription
  Interventions: Other: Pharmacist prescription
- Clinician prescription
  Interventions: Other: Clinician prescription

INTERVENTIONS:
Other: Pharmacist prescription — Pharmacist prescribed hormonal contraception (initiation or continuation).
  Groups: Pharmacist prescription
Other: Clinician prescription — Clinician prescribed hormonal contraception (initiation or continuation).
  Groups: Clinician prescription

SUMMARY:
Prospective cohort study of women presenting to initiate hormonal contraception, prescribed by a clinician or pharmacist. Women will be followed for one year to assess contraceptive continuation and unintended pregnancy rates, as well as measures of safety and acceptability.

DETAILED DESCRIPTION:
Direct prescription of hormonal contraception (HC) by pharmacists, without a doctor's visit or medical prescription, is a strategy to improve access to contraception and reduce unintended pregnancy. Oregon is the first state in the nation to implement legislation, as of January 1, 2016, expanding the scope of pharmacists to prescribe short-acting HCs. House Bill (HB) 2879 allows pharmacists to directly prescribe HC including the patch and pill, without a medical prescription. Women over 18 years of age can either initiate or continue HCs with a pharmacist, and women under 18 can continue a prescription.

This prospective cohort study of women presenting to initiate hormonal contraception, prescribed by a clinician or pharmacist, aims to determine contraceptive continuation and incident pregnancy rates between women receiving hormonal contraception from a pharmacist versus other prescriber. Women will be followed for one year to assess contraceptive continuation and unintended pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting to initiate hormonal contraception at a study pharmacy

Exclusion Criteria:

* Pregnancy
* Contraindications to hormonal contraception
* Under 18 years of age
* Unable or unwilling to consent

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women presenting to initiate hormonal contraception at a study pharmacy.
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2019-01-27 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Contraceptive continuation rates | 12 months
  Percentage of contraceptive continuation assessed through survey at 12 months among women who present for contraception in pharmacies.

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Rodriguez, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States